CLINICAL TRIAL: NCT02184520
Title: A Prospective Randomized Postmarket Clinical Study of the TRANSITION Stabilization System
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Globus Medical Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PS090007/A10
Record Dates: First submitted 2014-07-03; First posted 2014-07-09 (Estimated); Results first posted 2021-03-15 (Actual); Last update posted 2021-03-15 (Actual); Status verified 2021-02

CONDITIONS: Acute Instabilities Thoracic, Lumbar and Sacral Spine; Chronic Instabilities Thoracic, Lumbar and Sacral Spine; Deformities of the Thoracic, Lumbar and Sacral Spine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TRANSITION (Active Comparator): Stabilization System
  Interventions: Device: TRANSITION
- REVERE (Active Comparator): Stabilization System
  Interventions: Device: REVERE

INTERVENTIONS:
Device: TRANSITION
  Arms: TRANSITION
Device: REVERE
  Arms: REVERE

SUMMARY:
This postmarket surveillance study is being conducted to evaluate the TRANSITION Stabilization System as an adjunct to fusion in the treatment of acute or chronic instabilities or deformities of the thoracic, lumbar and sacral spine. The study will involve up to 360 subjects at no more than 20 sites, to be treated with the TRANSITION Stabilization System. The data from this postmarket surveillance study will be provided to FDA in accordance with the 522 order.

ELIGIBILITY:
Inclusion Criteria:

* Any of the following acute or chronic instabilities or deformities of the thoracic, lumbar or sacral spine:
* degenerative spondylolisthesis with objective evidence of neurologic impairment,
* kyphosis, or
* pseudoarthrosis (failed previous fusion)
* Age 18 or older at the time of consent
* Able to understand and sign informed consent form
* Psychosocially, mentally and physically able to comply with protocol
* Able to meet the proposed follow-up schedule at 6 mo, 12 mo, and 24 mo

Exclusion Criteria:

* Prior fusion surgery or another spinal device implanted in the thoracic, lumbar or sacral spine
* Requires treatment of more than two vertebral levels
* Lytic spondylolisthesis at the index level(s)
* Clinically compromised vertebral bodies at the affected level(s) due to current or past trauma
* Sustained pathologic fractures of the spine or hip, including prior fracture or trauma to vertebral structures at any thoracic, lumbar, or sacral level
* Morbid obesity defined as a body mass index > 40, or a weight more than 100 lbs over ideal body weight
* Pregnant or interested in becoming pregnant within the next 2 years
* Active systemic or local infection
* Known allergy to device materials titanium, polycarbonate (PCU), polyethylene terepthalate (PET), or hydroxyapatite (HA).
* Taking medications or any drug known to potentially interfere with bone/soft tissue healing (e.g., steroids, excluding routine NSAIDs)
* Systemic disease including AIDS, HIV, Hepatitis C
* Has an active malignancy defined as a history of any invasive malignancy (except non-melanoma skin cancer), unless he/she has been treated with curative intent and there has been no clinical signs or symptoms of the malignancy for at least 5 years
* Neuromuscular disorders such as muscular dystrophy, spinal muscular atrophy, amyotrophic lateral sclerosis, etc.
* Participation in an investigational device or drug clinical trials within 30 days of surgery
* Acute mental illness or substance abuse
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2016-04-19 (Actual); Primary Completion 2016-10-20 (Actual); Study Completion 2017-05-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Fort Wayne Orthopaedics, Fort Wayne, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study was terminated prior to primary and secondary endpoint data collection, therefore no study data is reported.
Groups:
- TRANSITION: Stabilization System
  TRANSITION
- REVERE: Stabilization System
  REVERE
Period: Overall Study
Arm/Group | TRANSITION | REVERE
Started | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The study was terminated prior to primary and secondary endpoint data collection, therefore no study data is reported.
Groups:
- Total: Total of all reporting groups
Arm/Group | TRANSITION | REVERE | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical
Age, Continuous
Sex: Female, Male
Race (NIH/OMB)

OUTCOME MEASURES:

1. Primary Outcome: Fusion Rates
Description: The study was terminated prior to primary and secondary endpoint data collection, therefore no study data is reported.
Time Frame: 24 months
Population: The study was terminated prior to primary and secondary endpoint data collection, therefore no study data is reported.
Arm/Group | TRANSITION | REVERE
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 24 months
Description: The study was terminated prior to primary and secondary endpoint data collection, therefore no study data is reported.
Arm/Group | TRANSITION | REVERE
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results.